CLINICAL TRIAL: NCT06356922
Title: Phase I/II Study Assessing Radioligand Therapy (RLT) Using [177Lu]Lu-PentixaTher for Relapsed/Refractory CXCR4+ Acute Leukemia.
Brief Title: Study Assessing RLT Using [177Lu]Lu-PentixaTher for Relapsed/Refractory CXCR4+ Acute Leukemia.
Acronym: PENTILULA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC20_0123
Record Dates: First submitted 2024-03-22; First posted 2024-04-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Acute Leukemia
MeSH Terms: interventions — Drugs, Investigational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [177Lu]Lu-PentixaTher (Experimental): Injection of [177Lu]Lu-PentixaTher
  Interventions: Drug: Experimental drug [177Lu]Lu-PentixaTher

INTERVENTIONS:
Drug: Experimental drug [177Lu]Lu-PentixaTher — Injection of [177Lu]Lu-PentixaTher

SUMMARY:
CXCR4 inhibition may represent a new therapeutic strategy in acute leukemia (AL) patients, not only by increasing chemosensitivity but also by preventing relapse of the disease by disruption of the interaction of residual leukemic cells with the bone marrow niche. Radiolabeled CXCR4 ligands have been developed for PET imaging (68Ga-PentixaFor; INN: Gallium (68Ga) boclatixafortide) and radioligand therapy (RLT) ([177Lu]Lu-PentixaTher/[90Y]Y-PentixaTher). [177Lu]Lu and [90Y]Y-PentixaTher have been tested in three multiple myeloma patients in named-patient use with a remarkable efficacy in 2 patients (Herrmann, 2016). Moreover, feasibility of CXCR4 PET imaging in AML was reported, providing a framework for future theranostic approaches targeting the CXCR4/CXCL12-defined leukemia-initiating cell niche (Herhaus, 2016).

Here a Phase I/II study to determine maximal tolerated dose (MTD) of a RLT using [177Lu]Lu-PentixaTher in relapsed/refractory AL was designed. This will be a standard phase I/II 3+3 dose escalation study. Five dose levels will be tested, so 6 to 21 patients have to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* AML/ALL (OMS) with >5% of blasts in bone marrow (with or without extramedullary localisation)
* CXCR4+ (ratio >2/isotypic control) at the time of pre-inclusion
* All previously treated AML/ALL patients who have experienced relapse or treatment failure with no alternative treatment
* At least 15 days since previous treatment
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Annex 6)
* eGFR ≥ 50 ml/min by MDRD or CKDEPI
* ASAT or ALAT > 5 upper normal value (except in case of documented presence of leukemia in the liver)
* Serum bilirubin ≤ 30 µmol/l
* Negative pregnancy test documented prior to enrolment (for females of childbearing potential)
* Agree to use an effective form of contraception with sexual partners throughout study participation (for female and male patients who are fertile)
* No active cardiac dysfunction (LVEF > 45%)
* DLCO >40%
* Written informed consent
* Be willing and able to comply with scheduled visits and study procedures
* Affiliation with French social security system or beneficiary from such system

Exclusion Criteria:

* Meningeal involvement
* HIV positive
* Active Hepatitis B or C
* Active infection within 7 days of starting treatment
* Previous or concurrent second malignancy except for adequately treated basal cell carcinoma of the skin, curatively treated in situ carcinoma of the cervix, curatively treated solid cancer, with no evidence of disease for at least 1 year
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
* Participation at the same time in another study in which investigational drugs are used
* Patient with contra-indications to Rhu-EPO, Rhu-GCSF, allopurinol, rasburicase, anti-histamines and corticosteroids
* Absence of written informed consent
* Pregnant or child breast feeding woman
* Patient under guardianship or trusteeship
* Patient under judicial protection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-10-22 (Estimated); Study Completion 2027-10-22 (Estimated)

PRIMARY OUTCOMES:
Safety of RLT using one injection of [177Lu]Lu-PentixaTher | Between Week 4 and Week 6
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Tolerance | Between Week 4 and Week 6
  Tolerance of the RLT will be evaluated by dosimetry studies, especially in terms of renal and hepatic doses delivered

SECONDARY OUTCOMES:
Overall response rate | Between Week 4 and Week 6
  Response evaluation (CR, CRp and PR) after the infusion of [177Lu]Lu-PentixaTher
Complete response rate | Between Week 4 and Week 6
  Response evaluation (CR, CRp) after the infusion of [177Lu]Lu-PentixaTher
Overall survival | Month 12
  Time interval from the date from initial of study treatment (D0) until the date of last follow-up or death
Leukemia-free survival | Month 12
  Time interval from the date of documented complete response (CR, CRp) until the date of last follow-up, death or relapse
Minimal residual disease | Month 12
  CXCR4 ratio by flow cytometry after [177Lu]Lu-PentixaTher
Whole-body biodistribution | Between Week 4 and Week 6
  Serial whole body scintigraphies
Plasma uptake | Between Week 4 and Week 6
  The activity in each plasma sample will be determined by counting 0,2 ml of plasma in a calibrated gamma counter with an appropriate window setting. The maximal uptake (%) and area under the curve (AUC) of [ 177Lu]Lu-PentixaTher at the target lesion, organs and blood will be determined
Radiation dosimetry | Between Week 4 and Week 6
  Whole body quantitative scintigraphies
Renal safety | Month 12
  Renal safety will be assessed by measuring creatinine
Renal safety | Month 12
  Renal safety will be assessed by measuring urea
Renal safety | Month 12
  Renal safety will be assessed by measuring eGFR by MDRD or CKDEPI
Renal safety | Month 12
  Renal safety will be assessed by measuring urinalysis
Correlation between different cytokines and toxicity | Month 12
  FLT3 and IL6 serum level
Factors associated response | Month 12
  Responses will be evaluated 4/6 weeks after the infusion of [177Lu]Lu-PentixaTher (Day 0): Complete remission (CR) is defined by normalization of the blood and the bone marrow with < or = 5% of blasts, neutrophil count > 1.109 /l and platelet count >100 Giga/l. CR with incomplete platelets recovery (CRp) is defined as for CR including platelet transfusion independence but with platelet count remaining below 100 Giga/l. Partial response (PR) is defined by blast clearance ≥50% in blood or bone marrow or bone marrow with > 5% and < 20 % of blasts
Exploratory outcome measure = Identification of biological biomarkers | Month 12
  Different cytokines including FLT3 and IL6 serum levels will be monitored by serial blood sampling at D1, D8, D15, D22 as well as during the monitoring visits at 1 month, and only FLT3 and IL6 at 3, 6, 9 and 12 months

OTHER OUTCOMES:
Predictive role of PET/MRI (ancillary study) | Between Week 4 and Week 6
  SUVmax will be recorded in extra-medullary sites of pathological uptake.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux, Gironde
  - CHU de Nantes, Nantes, Loire-Atlantique
  - CHU d'Angers, Angers, Maine et Loire
  - CHU de Clermont-Ferrand, Clermont-Ferrand, Puy de Dôme

IPD SHARING:
Plan to Share IPD: No